CLINICAL TRIAL: NCT04481542
Title: Aortic Dissection With 4-dimensional Phase-contrast Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019011776B0
Record Dates: First submitted 2020-02-23; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-03

CONDITIONS: MRI
Keywords: CVS MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: MRI — check MRI quality in aorta

SUMMARY:
We prospectively collected information on consecutive patients who had been evaluated using 4D PC-MRI for aortic pathology in a tertiary hospital between April 2018 and Feb 2020. Patients were eligible for inclusion in the study if they had a clinical indication for CTA of aortic dissections.

DETAILED DESCRIPTION:
The exclusion criteria were non-MRI-compatible ferromagnetic devices and pregnancy. In addition, patients with poor compliance and with unstable status that prevented them from lying down for the MRI protocol were excluded. Initially, 26 patients evaluated. One patient was excluded due to fever at the scheduled time, and another was unable to lie down due to complicated spine disease. All patients underwent CTA scan on a 64-slice multidetector scanner (Somatom Sensation 64; Siemens Healthcare, Erlangen, Germany) with the intravenous administration of contrast media, followed by 4D PC-MRI to assess aortic pathology

ELIGIBILITY:
Patients were eligible for inclusion in the study if they had a clinical indication for CTA of aortic dissections. The exclusion criteria were non-MRI-compatible ferromagnetic devices and pregnancy. In addition, patients with poor compliance and with unstable status that prevented them from lying down for the MRI protocol were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with aortic disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
stroke volume | 5 years
  anatomic/hemodynamic parameter

SECONDARY OUTCOMES:
adverse event | 5 years
  diagnostic function

CONTACTS AND LOCATIONS:
Locations (1):
- Yao-Kuang Huang, Chiayi City, Chiayi County, Taiwan

IPD SHARING:
Plan to Share IPD: No